CLINICAL TRIAL: NCT05669144
Title: Co-transplantation of Mesenchymal Stem Cell Derived Exosomes and Autologous Mitochondria for Patients Candidate for CABG Surgery With EF< 25% (Clinical Trial Phase ])
Brief Title: Co-transplantation of Mesenchymal Stem Cell Derived Exosomes and Autologous Mitochondria for Patients Candidate for CABG Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ahmadi tafti, professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.TUMS.THC.REC.1401.025
Record Dates: First submitted 2022-12-10; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Myocardial Infarction; Myocardial Ischemia; Myocardial Stunning
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia; Myocardial Stunning | interventions — Genes, Mitochondrial

STUDY DESIGN:
Intervention Model Description: 1. Intracoronary and intra-myocardial injection of exosomes (5 patients)
  2. Intracoronary and intra-myocardial injection of mitochondria (5 patients)
  3. Intracoronary and intra-myocardial injection of exosomes and mitochondria (5 patients)
  4. Placebo (5 patients)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- exosome therapy (Experimental): a) Intracoronary and intra-myocardial injection of exosomes (5 patients)
  1 mL of exosomes containing 100 micrograms of exosomes
  Interventions: Biological: mitochondria and MSC-derived exosomes
- mitochondria therapy (Experimental): b) Intracoronary and intra-myocardial injection of mitochondria (5 patients)
  1 mL of exosomes containing 10 million mitochondria
  Interventions: Biological: mitochondria and MSC-derived exosomes
- co-transplantation of mitochondria and exosome therapy (Experimental): c) co-transplantation Intracoronary and intra-myocardial injection of exosomes and mitochondria (5 patients)
  1 mL of exosomes containing 100 micrograms of exosomes
  1 mL of exosomes containing 10 million mitochondria
  Interventions: Biological: mitochondria and MSC-derived exosomes
- placebo (Placebo Comparator): 1 mL of placebo solution
  Interventions: Biological: mitochondria and MSC-derived exosomes

INTERVENTIONS:
Biological: mitochondria and MSC-derived exosomes — autologous mitochondria and MSC-derived exosomes

SUMMARY:
Heart failure (HF) and acute myocardial infarction that often follows are among the main causes of disability and death worldwide. As such, new treatments and biological drugs are needed to protect the heart against the harmful effects of ischemia and also reperfusion injury (IRI), preserve cardiac function, reduce the zone of myocardial infarction (MI), and improve patient outcomes. In this regard, it has been shown that mitochondrial dysfunction has a key role in the pathogenesis of heart ischemia, cardiomyopathy, and reperfusion injury. in this study which includes 4 groups of intervention, we try to minimize the damage by transplantation of mitochondria and administration of MSC-derived exosomes. MSC-derived exosomes limit inflammatory damage while fresh autologous exosomes limit oxidative stress.

DETAILED DESCRIPTION:
This research will be performed as a retrospective cohort study at Tehran Heart Center. Patients will be selected from CABG candidates with severely low Ejection fraction determined by speckle echocardiography. Patients with severe co-morbidities or cerebral damage will be excluded from the study. Detailed informed consent will be taken from the patients. Patients who refuse to provide consent will receive standard treatment.

Criteria

Inclusion Criteria:

* Patients who are a candidate for CABG due to CAD±MR
* History of Q-wave MI, less than one month
* Age: 35-80
* LVEF <=25% (by any imaging modality: echocardiography/SPECT/LV angiography and Cardiac MRI)
* Viability study as evidenced by low-dose dobutamine stress echocardiogram and/or thallium redistribution nuclear study (at least four viable segments).

Exclusion Criteria:

* Severe co-morbidities (e.g., renal failure, liver failure, etc.)
* Inability to provide informed consent
* Cerebral Damage

  1. Study groups:

     The standard treatment performed for all patients is revascularisation by coronary artery bypass grafting surgery. Patients will be divided into four groups based on the treatments received, in addition to the standard treatment.

     Mitochondrial and exosome transplantation by intracoronary and intra-myocardial injection. Study groups:
     1. Intracoronary and intra-myocardial injection of exosomes (5 patients)
     2. Intracoronary and intra-myocardial injection of mitochondria (5 patients)
     3. Intracoronary and intra-myocardial injection of exosomes and mitochondria (5 patients)
     4. Placebo (5 patients) For the patients in groups b and c, mitochondria will be extracted from a muscle tissue specimen extracted at the beginning of the surgery from pectoralis muscles exposed after sternotomy. Mitochondria will be extracted from the muscle specimen simultaneously with the surgery. When revascularisation is achieved by the bypass grafts, The extracted mitochondria will be injected into the heart muscle. A 31-gauge insulin syringe will perform injections into ten different sites in the ischemic area of the heart muscle. Besides direct injection into the heart muscle, one-third of the extracted mitochondria will be injected into the coronary sinus.

     Patients in groups a and b will receive the extracted exosome from MSC cells described in step 2. The extracted exosome will be injected into the coronary sinus after the placement of the Cardiopulmonary bypass.
  2. Isolation and characterisation of mesenchymal stem cells from the human umbilical cord (UC-MSCs) Human umbilical cord mesenchymal stem cells are enzymatically isolated by collagenase in terms of a previous study and cultured in DMEM / F12 medium with 10% exosome-depleted FBS (GMP grade) with penicillin and streptomycin antibiotics and incubated at 37 ° C and 5% CO2. After the cell confluence reaches 80%, the conditioned medium is collected (for exosome isolation, the cells are used in passage 3).

     The phenotypic analysis is performed on the third passage. Surface antigens are analysed for CD90, CD105, CD73 and CD34 using flow cytometry.
  3. Extraction of exosomes from UC-MSCs by ultracentrifugation and characterisation.

     After the cell confluence reaches 80%, the conditioned medium is collected for exosome isolation by several ultracentrifuges. In brief, after 48 h, the conditioned medium (CM) of the cells is centrifuged at 400 g for 10 min to remove cells and at 2500 g for 30 min to eliminate apoptotic bodies and debris. Afterwards, CM was centrifuged twice at 100 000 g for two h, followed by the process of suspending the exosome pellet in PBS.

     Surface antigens are analysed for CD9, CD63 and CD81 using western blot. Furthermore, Bradford Colorimetric Assay (BCA) kit is used to measure exosome production total protein at a wavelength of 570 nm. Dynamic light scattering (DLS) determines the size distribution of exosomes.
  4. Extraction of mitochondria from US-MSCs and characterisation.
  5. Short-term evaluation of the safety of clinical trial transplant mitochondria and exosome phase I:

     The patient will be under close monitoring after the surgery based on clinical symptoms, signs, arrhythmia, echocardiographic evaluations and lab results.
  6. Short-term evaluations of the patient in terms of blood factors (cTnT, CK-MB) Creatine kinase (CK) and its isoenzyme CK-MB are critical tools for diagnosing acute myocardial infarction (AMI). The content of CK-MB relative to total CK in myocardial cells is variable; in normal myocardium, it is low and enhanced several-fold in hypoxic myocardium and heart stroke.
  7. SPECT scan, Cardiac MRI and Dobutamine stress Speckle Echocardiography, before and after 2 months.

     The evaluation of the patient's recovery will be performed one month after the surgery. This evaluation is based on patients' signs and symptoms, Function Class assessments, Speckle and Dobutamine stress Eco, SPECT Nuclear heart Scan and Cardiac MRI imaging (CMR). Evaluations will be performed before surgery and one month after the surgery. Close Comparison will be performed between evaluation results to report possible improvements in the patient's condition.

     The assessed variables for follow-up evaluation include:
     * Ejection Fraction variables from Eco and CMR (LVEF, RVEF, Global EF)
     * 16 Segment viability analysis by SPECT scan and CMR
     * NYHA Classification assessment based on patient physical examination.
  8. Data Analysis will be performed by IBM SPSS Statistics Version 25. A p-value of less than 0.05 will be assessed as significant.

ELIGIBILITY:
Inclusion Criteria:

* • Patients who are candidate for CABG due to CAD±MR

  * History of Q-wave MI, less than one month
  * Age: 35-80
  * LVEF <=25% (by any imaging modality: echocardiography/SPECT/LV angiography and Cardiac MRI)
  * Viability study as evidenced by low-dose dobutamine stress echocardiogram and/or or thallium redistribution nuclear study (at least four viable segments).

Exclusion Criteria:

* Severe co-morbidities (e.g., renal failure, liver failure, etc.)

  * Inability to provide informed consent
  * Cerebral Damage

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-09-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
ejection fraction | 3 months
  left ventricle ejection fraction
allergic reactions | 3 months
  reactions including angioedema, hypotention, acute allergic reaction

SECONDARY OUTCOMES:
CK-MB | 2 week
  Creatine kinase (CK)
cTnT | 2 week
  cardiac troponin T
on pump duration | during the surgery
  on pump duration
ECMO duration | duration after surgery if needed
  extracorporeal membrane oxygenation duration
SPECT | 1 and 3 months post surgery
  defect size analysis
NYHA | 1 and 3 months post surgery
  cardiac function class
CMR | 1 and 3 months post surgery
  cardiac function

CONTACTS AND LOCATIONS:
Overall Officials: alireza hadizadeh, M.D, Study Chair — Tehran University of Medical Sciences
Locations (1):
- Tehran University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No